CLINICAL TRIAL: NCT00089882
Title: Risk Evaluation and Education for Alzheimer's Disease (REVEAL) II
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Robert C. Green, MD, MPH, Boston University
Other Study IDs: IA0057; 2R01HG002213-04 (NIH); Boston University SOM: H-23380
Record Dates: First submitted 2004-08-17; First posted 2004-08-18 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Apolipoproteins E (APOE); Genetic susceptibility testing
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: APOE Genetic susceptibility testing

SUMMARY:
The REVEAL II study provides healthy adult children and siblings of Alzheimer's disease patients with genetic testing and information about their own chances of developing the disease. The study will compare a condensed education and counseling program to the current more extensive program.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a common, progressive disease affecting memory and cognition. Apolipoprotein E (APOE) has been identified as a genetic factor that may increase the risk of developing Alzheimer's disease (AD). While several consensus statements have advised against the clinical use of APOE genotyping, each of these called for research to evaluate the impact of susceptibility genotyping and to explore the process of communicating about risk issues. The REVEAL I Study was funded in 1999 to enroll adult children of patients with AD to determine who would choose to obtain APOE genotyping, to devise an education and counseling protocol for the disclosure of APOE genotyping, and to study the impact of disclosing this information. The REVEAL I study demonstrated that Alzheimer's disease risk assessments with APOE genotyping can be given to relatives of people with Alzheimer's disease without causing severe adverse psychological or behavioral effects.

The REVEAL II study will examine whether receiving risk assessment and APOE genotyping disclosure through a Condensed Education and Counseling Protocol is as safe and as effective as receiving such information through our current Extended Protocol. This study will also examine whether there are any differences among groups who receive disclosure of APOE results and risk assessment by different provider types, such as a physician or a genetic counselor. At least one-third of the participants in REVEAL II will be African American, in order to explore how racial identity affects the desire to obtain genetic risk assessment and the impact of receiving it.

Individuals who have a parent or sibling affected by Alzheimer's disease may enter the study either by self-referral to the study coordinator or by recruitment. Participants will have a scheduled phone interview during which demographic information, their relative's medical history, attitudes toward genetic testing and risk assessment for Alzheimer's disease, and interest in going on to the next step of the study will be assessed. During the second step of the study, participants will be randomly assigned to one of three study arms. Participants in the control arm of the study will be given the full educational and counseling protocol as was originally developed in the first funding period of this study. All participants will have the opportunity to continue with the study and have their blood drawn for genotype analysis and risk assessment. Follow-up sessions will be provided with psychometric measures and questionnaires.

Participants will be seen by the genetic counselor for two follow-up appointments, six weeks and six months after disclosure of risk information. A final 12 month follow-up questionnaire will be completed by mail and will be followed by a phone call from the genetic counselor.

ELIGIBILITY:
Inclusion Criteria:

* Adult children or siblings of people with Alzheimer's disease.

Exclusion Criteria:

* Adult children or siblings of people with Alzheimer's disease who are unable to visit a study site.
* Persons with currently untreated depression, anxiety or severe mood disturbances.
* Persons with cognitive deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2003-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Green, MD, MPH, Principal Investigator — Boston University School of Medicine, Genetics Program and Alzheimer's Disease Center
Locations (4):
- United States (4):
  - Howard University College of Medicine, National Human Genome Center, Washington D.C., District of Columbia
  - Boston University School of Medicine, Alzheimer's Disease Center, Boston, Massachusetts
  - Weill Medical College of Cornell University, Memory Disorders Program, New York, New York
  - Case Western Reserve University, Memory and Aging Center, Cleveland, Ohio

REFERENCES:
- [Background] Hipps YG, Roberts JS, Farrer LA, Green RC. Differences between African Americans and Whites in their attitudes toward genetic testing for Alzheimer's disease. Genet Test. 2003 Spring;7(1):39-44. doi: 10.1089/109065703321560921. PMID 12820701
- [Background] Roberts JS, LaRusse SA, Katzen H, Whitehouse PJ, Barber M, Post SG, Relkin N, Quaid K, Pietrzak RH, Cupples LA, Farrer LA, Brown T, Green RC. Reasons for seeking genetic susceptibility testing among first-degree relatives of people with Alzheimer disease. Alzheimer Dis Assoc Disord. 2003 Apr-Jun;17(2):86-93. doi: 10.1097/00002093-200304000-00006. PMID 12794385
- [Background] Roberts JS, Barber M, Brown TM, Cupples LA, Farrer LA, LaRusse SA, Post SG, Quaid KA, Ravdin LD, Relkin NR, Sadovnick AD, Whitehouse PJ, Woodard JL, Green RC. Who seeks genetic susceptibility testing for Alzheimer's disease? Findings from a multisite, randomized clinical trial. Genet Med. 2004 Jul-Aug;6(4):197-203. doi: 10.1097/01.gim.0000132688.55591.77. PMID 15266207
- [Result] LaRusse S, Roberts JS, Marteau TM, Katzen H, Linnenbringer EL, Barber M, Whitehouse P, Quaid K, Brown T, Green RC, Relkin NR. Genetic susceptibility testing versus family history-based risk assessment: Impact on perceived risk of Alzheimer disease. Genet Med. 2005 Jan;7(1):48-53. doi: 10.1097/01.gim.0000151157.13716.6c. PMID 15654228
- [Result] Roberts JS, Cupples LA, Relkin NR, Whitehouse PJ, Green RC; REVEAL (Risk Evaluation and Education for Alzheimer's Disease) Study Group. Genetic risk assessment for adult children of people with Alzheimer's disease: the Risk Evaluation and Education for Alzheimer's Disease (REVEAL) study. J Geriatr Psychiatry Neurol. 2005 Dec;18(4):250-5. doi: 10.1177/0891988705281883. PMID 16306249
- [Derived] Christensen KD, Roberts JS, Zikmund-Fisher BJ, Kardia SL, McBride CM, Linnenbringer E, Green RC; REVEAL Study Group. Associations between self-referral and health behavior responses to genetic risk information. Genome Med. 2015 Jan 31;7(1):10. doi: 10.1186/s13073-014-0124-0. eCollection 2015. PMID 25642295